CLINICAL TRIAL: NCT03871920
Title: A Prospective Multi Center Prospective Cross-sectional and Longitudinal Study to Evaluate the Psychometric Properties of the Short Patient Evaluation Questionnaire
Brief Title: Psychometric Evaluation of the Short Patient Evaluation Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanco van der Maas (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); HES-SO Valais-Wallis (Other); University of Bern (Other)
Responsible Party: Sponsor-Investigator, Nanco van der Maas, Principle investigator, Institut fuer Physiotherapieforschung
Organization: Institut fuer Physiotherapieforschung (Other)
Other Study IDs: SPEQ
Record Dates: First submitted 2017-08-15; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Patient Reported Outcomes
Keywords: Physiotherapy; outcomes; therapy quality
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intervention: any kind of condition treated by physiotherapists, physical therapy treatment is chosen by treating physiotherapist
  Interventions: Other: physical therapy treatment

INTERVENTIONS:
Other: physical therapy treatment — any treatment chosen by treating physiotherapist

SUMMARY:
It is important for physiotherapy in general and for the individual physio-therapist to demonstrate the result of the interventions in physiotherapy. The new short (4 items) generic questionnaire Short Patient Evaluation Questionnaire SPEQ was especially developed for use in private practices to answer the main questions for evaluation of treatment. This research project aims at evaluating the reliability, validity and responsiveness of the SPEQ and at providing an estimate for Minimal Important Difference MID that may be used as threshold for clinical relevant changes.

DETAILED DESCRIPTION:
In this study the investigators evaluate the reliability, validity and responsiveness of the SPEQ and providing an estimate for Minimal Important Difference MID. They will use a longitudinal multicenter design with an adequate sample size of n=250 for validity and n=80 for reliability evaluation. Private practices and the Department of Physiotherapy of the Inselspital, Bern University Hospital, will participate in the study.

Reliability will be evaluated in a test-retest setting and with ordinal alpha. The SPEQ will be compared to the Euroqual-5-Dimensions-5-Levels (EQ-5D-5L), Short Form 12 (SF-12) and Patient Satisfaction Questionnaire (PSQ) to evaluate the validity. Responsiveness will be evaluated using a criterion validity approach and hypothesis testing of the correlation between SPEQ and the other questionnaires. In addition, the investigators will calculate ES, Standardized Response Mean (SRM), Modified SRM (MSRM) and relative efficiency between SPEQ and the criterions. For MID estimates, they use a combined anchor and distribution based approach. The anchors for the items are provided by the T0- and T1-questionnaire.

Patients will be recruited by the treating physiotherapists and provide written informed consent. At baseline, they will complete the T0-questionnaire, SF-12 and EQ-5D-5L. At the end of treatment or after 6 month of treatment for persons in long term treatment, the patients will fill out SPEQ, the T1-questionnaire, SF-12, EQ-5D-5L, and the PSQ. Two to seven days after the second test series, a subset of patients(n=80) will be asked to answer the SPEQ questions again by telephone.

Descriptive statistics will describe missing data, distribution of data over scale levels, frequency, floor and ceiling effects. Scaling will be tested by comparing pearson and spearman correlations and effect size (ES) for ordinal data and for metric data. Independence will be evaluated with the Mann-Whitney U test. The assumptions for building a sum of score will be evaluated comparing and assessing the spearman correlations and a categorical principle component analysis of the matrix of the 4 items of the SPEQ.

The reliability will be evaluated. Correlations between the SPEQ and the criterions EQ-5D-5L, SF-12 and PSQ will demonstrate validity.

Responsiveness will be evaluated analyzing the correlations between SPEQ and criterion and hypothesis testing of change of scores (Cosmin). Furthermore we will calculate the several traditional statistics; Effect Size, Standardized Response Mean, Modified Standardized Response Mean and relative efficiency between SPEQ and the criterion; distribution based Minimal Important Change estimates will be calculated with 0.5 Standard Deviation, Standard Error Measurement and Minimal Detectable Change at the 95% confidence interval; the mean between T0 and T1 values are anchor-based MID estimates. The range of anchor and distribution based MIC estimates will be analysed by Receiver Operating Characteristics curves. The result of the analysis provides an estimate that will be compared to the MID estimate of the criterion validity approach. Finally the threshold for clinical relevant change for the items and the sum of scores of the SPEQ will be determined.

The investigators expect the SPEQ to be a reliable, valid and responsive patient rated outcome assessment that can be used in the evaluation of the results of physiotherapy treatment.

ELIGIBILITY:
Inclusion criteria

* Persons older than 18 years, that are in physical therapy treatment.
* Persons must be able to read and understand German.

Exclusion criteria

* Grave cognitive changes
* Bedridden patients
* Grave comorbidities that may interfere with the treatment with physical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of the regular patient in full age in physical therapy treatment without a grave other health problems, that may interfere with the result of the treatment with physiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Test Retest reliability of SPEQ | up to 30 weeks
  Intra-Class Correlation coefficient (using a two way random effects model)
Accuracy of the SPEQ | up to 30 weeks
  analysis of accuracy of SPEQ to detect patients who changed in transition question with ROC analysis
Criterion Validity | up to 30 weeks
  The validity will be assessed using hypothesis testing of correlations (between SPEQ and existing previously validated measures). The SPEQ has a sufficient criterion validity, if these correlations are at least moderate (rho>0.5)

SECONDARY OUTCOMES:
Inner consistancy | up to 30 weeks
  The inner consistency will be calculated with ordinal alpha.
Construct validity of the SPEQ | up to 30 weeks
  Categorial principle component analysis of SPEQ will be performed to asses the construct validity of the SPEQ.
Responsiveness of the SPEQ | up to 30 weeks
  Sensitivity to change will be evaluated using Effect Size, Standardized Mean, Modified standardized Mean and Relative efficiency.
Validity of the SPEQ as assessed using Spearman correlations with scores of other previously validated measures | up to 30 weeks
  The validity of the SPEQ was determined by calculating Spearman correlations between SPEQ and scores of previously validated measures (EQ-5D-5L, SF-12 and SPQ). Scores >0.6 were considered indicative of high validity.

OTHER OUTCOMES:
Smallest sum of the proportions of misclassification | up to 30 weeks
  By defining a cut-off value at the smallest sum of the proportions of misclassification, the investigators will define Minimal Important Difference
Distribution based Minimal Important Difference | up to 30 weeks
  MID is defined for all items and the sum of item scores as 0.5 Standard Deviation, Standard Error Measurement and Minimal Detectable Change at the 95% confidence interval
Anchor based Minimal Important Difference | up to 30 weeks
  MID is defined for item 2, 3 and the sum of items scores as the average change between T1 and T2 for the subset of patients with a minimal change as determined by the transition question.

CONTACTS AND LOCATIONS:
Overall Officials: Nico van der Maas, Principal Investigator — Institut für Physiotherapieforschung gmbh, Biel, Switzerland; Martin Verra, PHD, Principal Investigator — Institute of physiotherapy, Insel university hospital, Bern, Switzerland; Roger Hilfiger, MSc., Principal Investigator — HES-SO Valais/Wallis, Leukerbad, Switzerland; Angela Balsimann Schwarz, MSc., Principal Investigator — Bern university of applied sciences, Health professions

IPD SHARING:
Plan to Share IPD: No